CLINICAL TRIAL: NCT01081418
Title: Assertive Community Treatment (ACT) as Part of Integrated Care Versus Standard Care: a 12-month Trial in Patients With First- and Negatively Selected Multiple-episode Schizophrenia-spectrum Disorders Treated With Quetiapine IR
Brief Title: Assertive Community Treatment (ACT) in Schizophrenia Spectrum Disorders
Acronym: ACCESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Associate Professor Martin Lambert, Psychosis Centre, Department of Psychiatry and Psychotherapy, University Medical Center Hamburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number: 2005-001069-32
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, assertive community treatment, quetiapine
MeSH Terms: conditions — Schizophrenia | interventions — Community Mental Health Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard care (Experimental): Standard care comprised a treatment network consisting of open and closed inpatient wards, day-clinics, an outpatient centre, and eight private psychiatrists. Each patient was treated by a private psychiatrist or by a psychiatrist in the outpatient centre. Home visits were possible, but office visits were the general rule. Patients were allowed to use all treatment offers in the outpatient centre. Outside office hours, patients could refer themselves to the psychiatric hospital. Psychosocial treatments as supportive therapy, psychoeducation, psychotherapy, and family intervention were provided infrequently and in a less intensive and unsystematic way, and only in the minority of cases. This 'standard of care' definition is in accordance with other studies.
  Interventions: Behavioral: Assertive Community Treatment (ACT)

INTERVENTIONS:
Behavioral: Assertive Community Treatment (ACT) — ACT was structured and implemented according to guidelines of the Assertive Community Treatment Association (ACTA). Team members were highly educated psychosis experts consisting of a consultant psychiatrist, a psychiatrist, two psychologists, and a nurse, all of which received training in cognitive behavioral (CBT), dynamic, and/or family psychotherapy. Study participants could use all treatment options within the integrated care program such as psychoeducation groups, social skills training, family groups, motivational addiction therapy, meta-cognitive training etc.
  Other Names: Assertive Community Treatment, Schizophrenia

SUMMARY:
The study examined the 12-month effectiveness of continuous therapeutic assertive community treatment (ACT) as part of integrated care (IC) compared to standard care (SC) in a catchment area comparison design in patients with schizophrenia spectrum disorders (SSD) treated with quetiapine IR.

DETAILED DESCRIPTION:
Two catchment areas in Hamburg, Germany with similar population size and health care structures were assigned to offer 12-month ACT (& IC; Department of Psychiatry and Psychotherapy, University Medical Center Hamburg-Eppendorf) or SC (Asklepios Hospital, Department of Psychiatry and Psychotherapy) to 120 first-episode and negatively selected multiple-episode patients with SSD. Primary outcome was the time to Service Disengagement. Secondary outcomes comprised medication non-adherence, improvements of symptoms, functioning, quality of life, satisfaction with care from patients and relatives perspectives, and service use data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Met the diagnostic criteria of a first- or multiple episode of a schizophrenia spectrum disorders, i.e. schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, or psychotic disorder NOS
* New initiation or current treatment with quetiapine Immediate Release (IR)

Exclusion Criteria:

* Other psychotic disorders (e.g., due to medical condition)
* Mental retardation (IQ lower than 70 points)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Time to Service Disengagement | 12 months
  The primary outcome of the study was the time to service disengagement (SD). This primary aim was chosen because the assertive approach of ACT is to prevent service disengagement3 and because service disengagement is a major predictor for relapse and thereby poor long-term outcome.16,17 Service disengagement was present, if a patient repeatedly refuses further treatment despite several attempts of reengagement (phone calls of patient and family in both treatment arms and potentially home visits in the ACT group).

SECONDARY OUTCOMES:
Improvements of symptoms, functioning, quality of life, and satisfaction with care from patients and relatives perspectives | 12 months
  Secondary outcomes comprised medication non-adherence, improvements of symptoms, functioning, quality of life, and satisfaction with care from patients and relatives perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lambert, MD, Principal Investigator — Psychosis Centre, Department of Psychiatry and Psychotherapy, University Medical Center Hamburg
Locations (1):
- University Medical Center Hamburg, Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Karow A, Brettschneider C, Helmut Konig H, Correll CU, Schottle D, Ludecke D, Rohenkohl A, Ruppelt F, Kraft V, Gallinat J, Lambert M. Better care for less money: cost-effectiveness of integrated care in multi-episode patients with severe psychosis. Acta Psychiatr Scand. 2020 Mar;141(3):221-230. doi: 10.1111/acps.13139. Epub 2020 Jan 12. PMID 31814102
- [Derived] Karow A, Reimer J, Konig HH, Heider D, Bock T, Huber C, Schottle D, Meister K, Rietschel L, Ohm G, Schulz H, Naber D, Schimmelmann BG, Lambert M. Cost-effectiveness of 12-month therapeutic assertive community treatment as part of integrated care versus standard care in patients with schizophrenia treated with quetiapine immediate release (ACCESS trial). J Clin Psychiatry. 2012 Mar;73(3):e402-8. doi: 10.4088/JCP.11m06875. PMID 22490266
- [Derived] Lambert M, Bock T, Schottle D, Golks D, Meister K, Rietschel L, Bussopulos A, Frieling M, Schodlbauer M, Burlon M, Huber CG, Ohm G, Pakrasi M, Chirazi-Stark MS, Naber D, Schimmelmann BG. Assertive community treatment as part of integrated care versus standard care: a 12-month trial in patients with first- and multiple-episode schizophrenia spectrum disorders treated with quetiapine immediate release (ACCESS trial). J Clin Psychiatry. 2010 Oct;71(10):1313-23. doi: 10.4088/JCP.09m05113yel. Epub 2010 Mar 23. PMID 20361911